CLINICAL TRIAL: NCT05668559
Title: The Effects of rTMS on Postoperative Cognitive Function in Patients After Cardiac Surgery
Brief Title: Transcranial Magnetic Stimulation and Perioperative Neurocognitive Disorders
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Anshi Wu (Other)
Responsible Party: Sponsor-Investigator, Anshi Wu, Director of department of anesthesiology, Chaoyang Hospital, Beijing Chao Yang Hospital
Organization: Beijing Chao Yang Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20221205
Record Dates: First submitted 2022-12-06; First posted 2022-12-30 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-08

CONDITIONS: Postoperative Cognitive Dysfunction; Repetitive Transcranial Magnetic Stimulation
MeSH Terms: conditions — Postoperative Cognitive Complications | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active rTMS Group (Experimental): A stimulation set will be administered to each participant in the rTMS group with 15 sessions stimulation for total five days after surgery.
  Interventions: Procedure: repetitive transcranial magnetic stimulation
- Sham Stimulation Group (Sham Comparator): Patients randomly assigned to sham group will receive 15 sessions sham stimulation for total five days after surgery.
  Interventions: Procedure: Sham Stimulation

INTERVENTIONS:
Procedure: repetitive transcranial magnetic stimulation — The rTMS mode consists of a cluster stimulus delivered every 0.2 seconds (5 Hz), with each cluster stimulus consisting of three burst stimuli with a 50 Hz body frequency. The duration of a single stimulus was approximately 40 seconds, for a total of 600 pulses. Stimulation takes place bilaterally in the dorsolateral prefrontal cortex (DLPFC).
  All enrolled patient in the rTMS group will receive 1 set simulation per day with an intersession interval (ISI) of over 30 minutes on postoperative day 1 to 5 after the surgery.
  Arms: Active rTMS Group
Procedure: Sham Stimulation — Shaman stimulation uses the same protocol (600 pulses per session, 3 sessions per set, ISI≥30 min, 3 sets) with the coil set at 90 against the skull on postoperative day 1 to 5 after the surgery.
  Arms: Sham Stimulation Group

SUMMARY:
To investigate the impact of rTMS on the incidence of perioperative neurocognitive disorders in patients after after cardiac surgerysurgery. To explore the underlying mechanisms behind the efficacy.

DETAILED DESCRIPTION:
There is a relatively high incidence of perioperative neurocognitive disorders（PND） after surgeries, and the incidence is even higher in the geriatric population undergoing cardiac surgery. Nevertheless, there remains no effective medication or intervention been approved in PND. It has been shown that brain stimulation can improve cognitive function in mild cognitively impaired patients. However, the effects on cognitive function in PND remain uninvestigated.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age 18 years or older.
* 2. ASA class I - III, patients undergoing elective cardiac surgery(coronary artery bypass grafting, aortic or mitral valve surgery).
* 3. Sign the informed consent.
* 4. Able to complete follow-up visits.

Exclusion Criteria:

* 1. A history of psychopathology and/or taking medication.
* 2. Previous history of neurological disease.
* 3. Severe organic diseases.
* 4. RTMS contraindications (such as a history of epileptic seizures, metal implants near the head).
* 5. Having delirium, assessed by CAM, before surgery.
* 6. Participating in other clinical studies at the time of screening.
* 7. Having a cardiopulmonary arrest and cardiopulmonary resuscitation.
* 8. Having short-term second operation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
The incidence of PND on the postoperative day 30 | Within 30 days after surgery
  Incidence of PND on the postoperative day 7 and day 30 will be defined according to the MOCA and MMSE.

SECONDARY OUTCOMES:
Postoperative delirium incidence | Within 7 days after surgery
  Incidence of postoperative delirium on postoperative day 1 to 7 will be defined by the Confusion Assessment Method for The Intensive Care Unit (CAM-ICU) or CAM
Perioperative pain | Within 7 days after surgery
  This will be assessed by using Visual Analogue Scale (VAS). The patients scored according to the severity of their pain from no pain (0) to most painful (10).
Sleep quality | Within 30 days after surgery
  We will use the Pittsburgh Sleep Quality Index (PSQI) to evaluate sleep quality. PSQI uses a 19-item questionnaire to assess sleep quality over one month30. An increased score indicates poor quality sleep. PSQI will be recorded at different points of time as follows：
  1. 1 day before surgery
  2. 7 days after surgery
  3. 30 days after surgery
Depressive symptom | Within 7 days after surgery
  Depressive disorder and depression symptom severity will be measured using the 9-item patient health questionnaire (PHQ-9). It is self-administered and carries a score ranging from 0 to 27, with a score range of 0 to 3. Five, ten, fifteen, and twenty are the thresholds for mild, moderate, and moderately severe depression.
Activities of daily living（ADL） | Within 30 days after surgery
  As part of the pre-surgery and post-surgery evaluations, the Chinese version of the ADL scale will be used, including a Physical Self-Maintenance Scale and an Instrumental ADL scale. ADL consists of 14 items, and the total score ranges between 14 and 56 points, with higher scores indicating a lower level of functioning. ADL will be evaluated at different points of time as follows：
  1. 1 day before surgery
  2. 7 days after surgery
  3. 30 days after surgery
Length of hospital stay | From the date of admission until discharged from hospital, up to 30 days
  A hospital length of stay is the number of days the patient spends in the hospital following surgery.
Length of ICU stay | From the date of admission until discharged from ICU, up to 30 days
  Similarly, the ICU length of stay was defined as the number of days the patient spent in the ICU before transferring to a general inpatient cardiac surgery ward
EEG characteristics | Within 30 days after surgery
  Electroencephalography will be recorded at different points of time as follows and EEG characteristics including power in alpha, beta, theta, delta, gamma, spectrum will be extracted using MATLAB. In addition, functional brain connectivity and brain network will be assessed at different points of time as follows：
  1. before anesthesia introduction
  2. during anesthesia
  3. on the 1th dayday after surgery
  4. on the 7th day after surgery
  5. on the 30th day after surgery
Incidence of major adverse cardiac and cerebral events | Within 30 days after surgery
  MACCE comprises all-cause mortality, myocardial infarction, repeat unplanned revascularization (surgical revision or percutaneous transluminal coronary angioplasty), and stroke

CONTACTS AND LOCATIONS:
Overall Officials: Anshi Wu, Study Director — Beijing Chao Yang Hospital

REFERENCES:
- [Derived] Wang J, Wang X, Li S, Yang J, Yan X, Gao J, Jia X, Zuo L, Wu A, Wei C. The effect of repetitive transcranial magnetic stimulation (rTMS) on perioperative neurocognitive disorders in patients after cardiac surgery: study protocol for a randomized controlled trial. Trials. 2025 Jul 24;26(1):253. doi: 10.1186/s13063-025-08988-3. PMID 40707956